CLINICAL TRIAL: NCT03238313
Title: Evaluation of "Plan A" Video Intervention
Brief Title: Evaluation of "Plan A"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: The Office of Adolescent Health, HHS (U.S. Federal Agency); Sentient Research (Industry); Planned Parenthood Mar Monte (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TP2AH000036
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plan A (Experimental): Plan A is the treatment condition. It is a 23-minute video that is designed to promote effective contraceptive use, use of dual methods of protection (condom use and prescription birth control use), and HIV/STI testing in African/American and Latina young women.
  Interventions: Behavioral: Plan A
- Toxic Life Cycle of a Cigarette (Active Comparator): The Toxic Life Cycle of a Cigarette is the counterfactual condition. It is a 17-minute video, but contains no information about reproductive health. Instead, the video teaches about the harms of cigarettes.
  Interventions: Behavioral: Toxic Life Cycle of a Cigarette

INTERVENTIONS:
Behavioral: Plan A
  Arms: Plan A
Behavioral: Toxic Life Cycle of a Cigarette — Video
  Arms: Toxic Life Cycle of a Cigarette

SUMMARY:
The purpose of the study is to determine if exposure to the "Plan A" video influences viewers' uptake of LARC, reduces unprotected sexual activity, and increases receipt of STI testing.

DETAILED DESCRIPTION:
The Policy & Research Group (PRG) is evaluating the "Plan A" video, which was designed to promote effective contraceptive use, use of dual methods of protection (condom use and prescription birth control use), and HIV/STI testing in African/American and Latina young women. The video is approximately 23 minutes in length and is shown immediately prior to a clinical appointment at a reproductive health center. By delivering the intervention prior to a clinic appointment, developers hope to reach high-risk teens at a teachable moment, when they can ask a health care provider about what they have learned. The primary focus of the study is to investigate the impact of the intervention on participants': 1) LARC use; 2) times having sex without a condom; and 3) STI testing. Secondary outcome measures include assessing the impact of the intervention on participants': 1) use of dual methods of protection during vaginal sex; and 2) use of other effective contraceptive methods. Finally, the evaluation will include exploratory analysis of participants': 1) perception of risk and/or severity for pregnancy and HIV/STI infection; (2) intention to use LARC; (3) intention to use other effective contraception methods; (4) provider communication self-efficacy; (5) condom negotiation self-efficacy; and (6) knowledge/awareness of contraception options/LARC.

The control (counterfactual) condition consists of a 17-minute video titled "The Toxic Life Cycle of a Cigarette". The control video, which discusses the effects of smoking, is shown in the same manner as the treatment video: immediately prior to a clinic appointment at a reproductive health center.

All eligible participants who provide the proper consent are randomized and enrolled into the study by a study coordinator who is an employee of the reproductive health clinic. Outcomes will be assessed using self-reported, participant-level data gathered (by way of a questionnaire) at three time points: baseline (enrollment, prior to watching the video); 3-month follow-up (3 months after baseline); and 9-month follow-up (9 months after baseline). The study is taking place at seven clinics within the Planned Parenthood Mar Monte system in California, all of which serve the target population.

ELIGIBILITY:
Inclusion Criteria:

* Be female
* Be 18 or 19 years old
* Self-identify as Latina and/or African-American
* Be visiting a reproductive healthcare provider at the study site
* Be deemed appropriate for the study by study staff/clinic staff with regards to physical and mental health and capacity
* Consent to participate in the study

Exclusion Criteria:

* Knowingly pregnant
* Trying to become pregnant
* Previously enrolled in the study
* Enrolled in studies in the same geographic area that aim to prevent teen pregnancy

Ages: 18 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — To be eligible to participate in the study, participants must self-report that they identify as 'female' when given the following list of options: Female; Male; Transgender; Do not identify as female, male, or transgender; Unknown
Enrollment: 1770 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
LARC Use | Three months after intervention
  Participant self-report on the use of Long Acting Reversible Contraception (LARC). Measured through one survey question which asks the participant to select all methods of prescription birth control currently being used.
STI Testing | Three months after intervention
  Participant self-report on if they have been tested for Sexually Transmitted Infections (STIs). Measured through two survey questions which ask the participant about whether they have ever been tested for STIs and if yes, whether they have been tested for STIs (other than HIV) in the past three months.
Times Having Sex Without a Condom | Three months after intervention
  Participant self-report on the number of times they have had vaginal, oral, or anal sex without a condom in the last three months. Measured through three survey questions which ask the participant how many times they have had vaginal, oral, and anal sex in the past three months.

SECONDARY OUTCOMES:
Use of Other Effective Contraception | Three months after intervention
  Participant self-report on the use of other effective contraceptive methods (oral contraceptives, patch, ring, and shot/injection). Measured through one survey question which asks the participant to select all methods of prescription birth control currently being used.
Dual Methods of Contraception | Three months after intervention
  Participant self-report on the use of dual methods of contraception (using a condom and another prescription birth control). Measured through two survey questions which ask participants how many times they have had vaginal sex in the past three months and how many times, of the times they had vaginal sex in the past three months, did they use both a condom and a form of prescription birth control.

OTHER OUTCOMES:
Perceived Risk of Pregnancy | Three months after intervention
  Participant self-report on perceived risk and severity of becoming pregnant and acquiring sexually transmitted infections or HIV. Measured through four survey questions which ask participants to rate their likelihood of becoming pregnant and acquiring HIV and STIs given various risky behaviors.
Intention to Use LARC | Three months after intervention
  Participant self-report on intention to use LARC. Measured through one survey question which asks participants to indicate how likely they are to use LARC in the next year.
Intention to Use Other Effective Contraception Methods | Three months after intervention
  Participant self-report on intention to use other effective contraception. Measured through two survey questions which asks participants to indicate how likely they are to use short-acting and long-acting prescription birth control in the next year.
Provider Communication Self-efficacy | Three months after intervention
  Participant self-report on perceived confidence in being able to communicate with health care providers. Measured through five survey questions where participants are asked to indicate their confidence level with talking to and receiving information from a health care provider.
Condom Negotiation Self-efficacy | Three months after intervention
  Participant self-report on perceived confidence in being able to negotiate condom use with her partner during sex. Measured through four survey questions which ask participants to report their level of confidence in discussing and using condoms with their partners.
Knowledge and Awareness of Contraception Options/LARC | Three months after intervention
  Participant self-report on knowledge and awareness of contraceptive options. Measured through 10 survey questions which ask participants to answer True/False questions about various kinds of contraception.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jenner, PhD, MMC, BA, Principal Investigator — The Policy & Research Group
Locations (1):
- The Policy & Research Group, Multiple Locations, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A dataset will be prepared at the conclusion of the study, which includes de-identified individual-level data on all study participants who contributed self-report data. Respondents will be represented only by a research ID number. Included in the dataset will be self-report data collected across all survey administrations (including demographic characteristics, sexual behaviors, and theoretical antecedents to those behaviors) and select information on program participation (e.g., which program sessions were attended). Basic data cleaning steps will be taken in order to ensure data are unidentifiable and to increase usability.
Time Frame: The individual participant dataset will become available twelve months after the study has concluded.

REFERENCES:
- [Derived] Jenner E, Walsh S, Henley C, Demby H, Leger R, Falk G. Randomized Trial of a Sexual Health Video Intervention for Black and Hispanic Adolescent Females. Prev Sci. 2023 Dec;24(Suppl 2):262-271. doi: 10.1007/s11121-023-01499-0. Epub 2023 Feb 3. PMID 36735143
- Available data/document: Information on publicly available dataset — https://documentcloud.adobe.com/link/review?uri=urn:aaid:scds:US:a6e30fe6-fb70-4d4a-9ab5-7a98da6084bb — For any individuals interested in accessing a copy of this public use dataset, please email info@policyandresearch.com with your inquiry.

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT03238313/SAP_000.pdf